CLINICAL TRIAL: NCT05212688
Title: A Randomised Phase II Study to Investigate the Effectiveness of ACUpuncture for the Relief of Long COVID Related Fatigue.
Brief Title: Randomised Study to Investigate the Effectiveness of Acupuncture for the Relief of Long COVID-19 Related Fatigue
Acronym: ACU-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCR5576
Record Dates: First submitted 2022-01-26; First posted 2022-01-28 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Acupuncture vs Control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Active Comparator): * Weekly treatment of 15 minutes for 6 weeks using Seirin 36 g 30 mm needles applied to two upper midline sternal points, thoracic paravertebral points, 5 pairs, 2 bilateral Trapezius trigger points, LI4, TE5, ST36, GB34, SP6, LR3 bilaterally, GV20 & GV24 midline
  * A maximum of two upper sternal indwelling studs [Seirin Pyonex semi-permanent studs] may be used after the second treatment if dyspnoea is present
  * Instructions will be given to massage the studs for 1 minute prior to exercise, if dyspnoeic or if very anxious, as often as necessary up to 12 times/day
  * Patients will be asked to rest for 15 minutes after each acupuncture treatment.
  * Clear instructions about self-needling for ongoing maintenance will be given to each patient
  The acupuncture will be given in 6 sessions at weekly intervals. Delays of up to 2 weeks in delivery of acupuncture are allowed within the protocol. The timing of the study questionnaires at weeks 2, 6 and 12 will remain unchanged.
  Interventions: Other: Acupuncture
- Active Control (Active Comparator): Patients randomised to the Active Control will be contacted once per week for 6 weeks for a semi-structured telephone consultation. Delays of up to 2 weeks in delivery of the Active Control session are allowed within the protocol. Patients will be asked during the telephone call to complete the study questionnaires at week 0, 2, 6. Participants will also be asked after the telephone call to rest for 15 minutes if they are able. The patients will also be telephoned on week 12 to complete the study assessments. Patients in Arm B will be required to attend RM in person for the baseline visit and at week 6 to perform the 1 Minute Sit to Stand Test (1-MSTS). The 1-MSTS can be performed virtually rather than in person. Other visits will be telephone calls and completion of questionnaires (paper or via patient portal) Once patients in the Active Control group have completed the 12 week study assessments, they will be offered crossover to receive acupuncture.
  Interventions: Other: Active Control

INTERVENTIONS:
Other: Acupuncture — Weekly treatment of 15 minutes for 6 weeks using Seirin 36 g 30 mm needles applied to two upper midline sternal points, thoracic paravertebral points, 5 pairs, 2 bilateral Trapezius trigger points, LI4, TE5, ST36, GB34, SP6, LR3 bilaterally, GV20 & GV24 midline.
  Arms: Acupuncture
Other: Active Control — Weekly contact once per week for 6 weeks for a semi-structured telephone consultation.
  Arms: Active Control

SUMMARY:
The Covid pandemic has left us with a significant number of people suffering from Long COVID, which is a clinical diagnosis of significant and varying ongoing symptoms at least 12 weeks following COVID-19 infection and characterised frequently by fatigue and breathlessness. Acupuncture has been shown to help breathlessness and fatigue in other conditions including in patients with cancer. Cancer related fatigue in the largest study, was assessed by the multiple functional inventory (MFI) score, assessing 5 domains of health, to give a single score.

We aim to randomise 160 patients, 80 in each arm. Randomisation and recruitment should take 24 months.

Each patient will be offered 6 weeks of weekly acupuncture treatment with a structured questionnaire on wellbeing or no acupuncture with a structure questionnaire on well-being. Both groups of patients will be given continued general advice on management of their symptoms. The next point of involvement will be at 12 weeks which will also be the final visit unless patients in Arm B (Active Control) chose crossover to receive acupuncture. Data at this point will correspond to the end of the participants participation. Over the next 3 months data will be cleaned and analysed.

The primary endpoint is General Fatigue scores, as self-reported by patients using the MFI, at 6 weeks. A 2-unit difference between groups (Acupuncture vs Active Control) in General Fatigue score is considered clinically important.

The secondary endpoints will include differences in scores of various questionnaires and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent.
2. Male or female, age > 18 years.
3. Female patients of childbearing age must confirm their intention not to fall pregnant during the study period of 6 weeks.
4. A clinical diagnosis of Long COVID a fatigue score of ≥ 5 on the C19-YRS First Assessment
5. A self-reported fatigue score on the C19-YRS ≥ 2 points more severe than their pre-COVID baseline
6. More than 12 weeks following a positive COVID-19 swab test (lateral flow or PCR) or an illness in keeping with COVID-19 infection in the opinion of the Chief Investigator, despite the absence of swab confirmation (not tested or test negative).
7. Where applicable, have completed any other therapeutic rehabilitation intervention for Long COVID-related fatigue.
8. Willing and able to attend for a course of 6 once per week acupuncture treatments
9. Co-existing reversible causes of fatigue and/or breathlessness medically optimized
10. If a patient has ongoing breathlessness a chest X-ray should have been performed
11. If on steroids should be on stable dose for at least two weeks at time of study entry
12. If taking other dietary/vitamin interventions should be on a stable regimen for at least two weeks at the time of study entry
13. If vaccinated should be a least two weeks post last vaccine dose or booster
14. Participants with a history of cancer must be on a stable dose of treatments such as oral TKIs, or antiestrogen therapies or be more than 2 years from diagnosis and completion of radical treatment
15. Where applicable, participants on aspirin, clopidogrel or oral anticoagulants are on a stable dose and discussed with the acupuncture clinician (Dr Jacqueline Filshie or a suitably qualified member of her team) before study entry.

Exclusion Criteria:

1. Recent acupuncture in the last 4 weeks
2. Contraindication to acupuncture in the opinion of the acupuncture clinician (Dr Jacqueline Filshie or a suitably qualified member of her team).
3. Patients currently receiving chemotherapy or immunotherapy at regular intervals likely to induce cyclical fatigue or within the last 12 months.
4. Patients currently receiving radiotherapy or within the last 12 months
5. Pregnancy
6. Patients with heart valve pathology/dysfunction are contra-indicated from using semi-permanent acupuncture studs for maintenance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
General Fatigue Score | 6 weeks
  The primary outcome will be the difference in General Fatigue scores, as self-reported by patients using the MFI ( Multidimensional Fatigue Inventory)
  , at 6 weeks. The MFI is a brief 20 item validated scale measuring general fatigue and other dimensions of physical and mental fatigue, activity and motivation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No